CLINICAL TRIAL: NCT03751423
Title: Intravenous Ketamine for Pain Control During First Trimester Surgical Abortion
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study on-hold due to COVID-19 pandemic restrictions. Will resume when possible.
Sponsor: Dr. Marie Eve Sophie Bussiere-Cote (Other)
Responsible Party: Sponsor-Investigator, Dr. Marie Eve Sophie Bussiere-Cote, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OBGY-KET-18
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Abortion in First Trimester
Keywords: procedural sedation; ketamine; fentanyl; morphine
MeSH Terms: interventions — Morphine; Fentanyl; Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, controlled, double-blinded, single-centre superiority trial with three parallel groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For the three treatment arms, the nurses, the study participants, and the abortion provider will be blinded to study arm assignment and will remain blinded throughout the course of the study. As such, all study personnel who will be administering questionnaires will be appropriately blinded to minimize bias. The provider of the IV medications will not be blinded. This decision was made in order to ensure participant safety in titrating medication doses, and to avoid the need to unblind all members if a reversal agent is required. The provider of the anesthetic will not disclose which study arm the participant belongs to and will not be involved in administering questionnaires or data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PO Morphine & IV Placebo (Active Comparator): One third of study participants will be randomized to this local standard of care arm.
  Interventions: Drug: PO Morphine; Drug: IV Placebo
- IV Fentanyl & PO Placebo (Active Comparator): One third of study participants will be randomized to this current gold standard of care arm.
  Interventions: Drug: IV Fentanyl; Drug: PO Placebo
- IV Ketamine & PO Placebo (Experimental): One third of study participants will be randomized to this experimental arm.
  Interventions: Drug: IV Ketamine; Drug: PO Placebo

INTERVENTIONS:
Drug: PO Morphine — 10-20mg oral morphine depending on such factors as weight (100-200mcg/kg), previous opiate exposure (opiate naïve vs opiate sensitized), and participant's previous experiences with opiate medications for painful procedures. Dosing will be determined at the discretion of the surgical provider in clinic that day, as per standard of care.
  Other Names: Morphine Sulphate
  Arms: PO Morphine & IV Placebo
Drug: IV Fentanyl — 0.5-1mcg/kg IV fentanyl over 2 minutes repeated every 5 minutes as needed until appropriate analgesia is reached.
  Other Names: Fentanyl Citrate Injection
  Arms: IV Fentanyl & PO Placebo
Drug: IV Ketamine — 200-500mcg/kg IV over 2 minutes repeated every 5 minutes as needed until appropriate analgesia is reached
  Other Names: Ketamine Hydrochloride Injection
  Arms: IV Ketamine & PO Placebo
Drug: PO Placebo — A standard placebo pill, the same size, shape and colour of the oral morphine. The placebo will be administered to the participants randomized to the IV ketamine and IV fentanyl during pre-op in the same manner the oral morphine would be administered.
  Other Names: Oral Placebo Pill
  Arms: IV Fentanyl & PO Placebo; IV Ketamine & PO Placebo
Drug: IV Placebo — This normal saline will be administered to the participants randomized to the oral morphine group during the procedure in the same manner that IV fentanyl or IV ketamine would be administered.
  Other Names: Normal Saline
  Arms: PO Morphine & IV Placebo

SUMMARY:
A therapeutic abortion is one of the most common procedures performed in Canada, with approximately 100,000 occurring annually. 95% of induced abortions are done surgically, with just over two thirds of these procedures taking place in the first trimester.

This study will be a randomized, controlled, double-blinded, single-centre superiority trial with three parallel groups; oral morphine vs intravenous fentanyl vs intravenous ketamine. The primary outcome will be immediate post-operative pain following a first trimester therapeutic abortion as assessed using the visual analogue scale. Randomization will be performed as block randomization with a 1:1:1 allocation ratio. In total, 123 participants will be recruited and randomized, with 41 being assigned to each treatment arm. This study will be conducted at the Women's Clinic at Kingston General Hospital in Kingston, Ontario, Canada. Women from Kingston and the surrounding areas are referred to this clinic and can self-refer for therapeutic abortion.

The investogators hope that this research will move us towards a better form of pain control for our participants undergoing first trimester surgical abortion, without increasing length of stay, side effects, or adverse events. This, in turn, will hopefully improve access to optimal pain control to participants undergoing first trimester surgical abortion in an outpatient setting.

DETAILED DESCRIPTION:
Rationale:

At present, the gold standard for pain control during first trimester abortion is the combination of a paracervical block with moderate intravenous (IV) sedation. Paracervical blocks are routinely done with lidocaine, with or without epinephrine or vasopressin. Moderate sedation is commonly achieved using fentanyl 50-100ug IV and midazolam 1-2mg IV. The issue with the use of IV opioids for sedation is the need for continuous cardio-respiratory monitoring, due to the risk of cardio-respiratory depression or collapse. This therefore limits the ability of some centers to provide the best form of pain control for their participants undergoing first trimester surgical abortion. For instance, our center currently uses a paracervical block plus a combination of oral medications (morphine and lorazepam), which has been found to be inferior to a paracervical block plus IV sedation. All participants without contraindications to NSAIDs are pre-medicated with naproxen as recommended.2 The investigators also have access to nitrous oxide/oxygen 50:50 (Entonox) to use as an adjunct, however this has not been found to significantly improve procedural or post-operative pain.

In the past, ketamine was used for pain control during first trimester abortion. Ketamine is a dissociative agent and does not carry the same risk of cardio-respiratory depression as intravenous opioids. Ketamine was felt to be ideal for first trimester surgical abortion -as the medication has uterotonic properties, which could result in less blood loss. Doses of 0.5mg/kg IV were typically used. However, the use of ketamine for first trimester surgical abortion decreased dramatically after the 1970-1980's due to reports of adverse events including emergence phenomena (nightmares), nausea, and vomiting. In fact, only one study published during this time did not find negative emergence phenomena in participants exposed to ketamine. More recently, a systematic review concluded that ketamine was an inferior agent when compared to propofol for pain control during first trimester surgical abortion. However, propofol, a general anesthetic requiring continuous cardio-respiratory monitoring, should not be placed in the same anesthetic category as ketamine. Furthermore, propofol is only available in a limited number of settings offering first trimester surgical abortion.

Over the last 10 to 15 years, ketamine has become an increasingly commonly used dissociative agent for procedural sedation in the emergency department. The benefits of its use include the simultaneous provision of both sedation and analgesia, while maintaining airway reflexes and respiratory drive. Intravenous ketamine use in the emergency department has been shown to yield high success rates (94% to 100%). In addition, of all the drugs commonly used in this setting, ketamine has one of the highest safety profiles and lowest rates of complications.

The investigators are interested in re-visiting whether ketamine would be an appropriate choice of anesthetic for first trimester surgical abortion. If ketamine is found to be superior to IV fentanyl, it would potentially increase access to optimal pain control in settings where continuous cardio-respiratory monitoring is not available. Furthermore, in the current era of opioid misuse, it is important that providers look for alternative forms of pain management when appropriate. In fact, the Society for Family Planning recently put out a call to action for more research on alternative options to control pain short of moderate or deep sedation.

Study Setting:

This study will be conducted at the Women's Clinic at Kingston General Hospital in Kingston, Ontario, Canada. Women from Kingston and the surrounding areas are referred to this clinic and can self-refer for therapeutic abortion.

Study Drugs:

* PO Morphine
* IV Fentanyl
* IV Ketamine
* PO Placebo
* IV Placebo

Administration of Study Drugs:

Once written informed consent is received the care provider will determine opiate sensitization stratum and write orders for the appropriate amount of oral morphine to be dispensed to the participant.

The next sequential randomization envelope for the appropriate stratum will then be retrieved. Within the randomization envelope there will be two envelopes, one for nursing staff and one for the anesthetist. Drug dispensing will be done in two stages.

Nursing staff will open their envelope to determine from which drawer they are to dispense the oral morphine dose ordered by the care provider (A, B or C). Two will be placebo and one will be oral morphine, but nursing staff will be blinded to group assignment.

The anesthetist will open her envelope prior to the procedure to determine group assignment. She will be responsible for the mixing and administration of all IV medications and will not be blinded to group assignment. All other study staff, clinical staff and the participant will remain blinded to group assignment.

Nursing staff will be responsible for dispensing and administering all other standard medications including dimenhydrinate, naproxen, lorazepam and misoprostol.

For all participants the anesthetist will prepare IV medications according to participant group assignment, ketamine, fentanyl or normal saline only. The syringes will be labelled with the participant's name and hospital identification number. The syringes will be used for IV drug administration during the procedure. Naloxone and/or midazolam will be administered as needed at the discretion of the anesthetist.

Standard Script:

Prior to starting the procedure, the physician administrating sedation during the procedure will inquire into some of the participant's favorite places and/or ideas, as this will be used to individualize guided imagery for each participant during the procedure. An example of such guided imagery during the procedure may include the physician asking the participant to feel the sand on her feet at her favorite beach, to hear the waves landing on the shore, and to feel the warmth of the sun on her skin. In addition to guided imagery performed during the procedure, the voices in the room will be minimized only to necessary communication in a calm gentle tone, and soothing music will be played quietly in the background. The guided imagery and room setup will be used for all participants, regardless of the study drug that they receive.

Consent Process:

Once the participant registers at the Women's Clinic, she will be asked by the nurse at intake if she would be interested in participating in the research study. If she is agreeable, the surgeon will proceed with the consent process.

If the participant consents to participate in the study, the surgeon will administer a questionnaire to obtain a thorough medical history, collect information on participant demographics and determine whether the participant is opiate naïve or opiate sensitized.

Randomization:

Participants will be randomized to one of three treatment arms following receipt of written informed consent.

Allocation Sequence Generation:

The allocation sequence will be generated by an epidemiologist in the Department of Obstetrics and Gynecology at Queen's University. Randomization will be blocked and stratified. Stratification will be based on the participant's current opiate usage to ensure that participants who are opiate sensitized are evenly distributed between the groups. Unique allocation sequences will be generated for each stratum. Random block sizes of 3 and 6 will be used for each of the sequences. For both sequences, participants will be allocated in a 1:1:1 ratio, with equal chance of being assigned to all three groups. An appropriate statistical program will be used to generate the two allocation sequences.

Randomization Process:

Randomization will be done with consecutively numbered opaque envelopes. Research staff will assemble these envelopes based on the two allocation sequences. The envelopes will be clearly labelled with the stratum (opiate sensitized or naïve). Within each envelope there will be two envelopes, one for nursing staff and one for the anesthetist. A sheet within the envelope for the nursing staff will indicate from which drawer they are to dispense the oral morphine (A, B, C). This will be done to ensure that nursing staff remains blinded to group assignment. A sheet inside the envelope for the anesthetist will indicate arm allocation (PO morphine, IV ketamine, IV fentanyl). The envelopes and sheets will be identical, except for the number and strata label on the outside and text on the sheet inside, to minimize the chance of accidental unblinding.

Upon receipt of written informed consent, the care provider will determine whether the participant is opiate sensitized or naïve and write an order for an oral morphine dose. The participant will be randomized by selecting the next envelope in the sequence of the appropriate stratum based on the consecutive numbering. Nursing staff will open their labeled envelope to determine from where to dispense the oral morphine. The anesthetist will open her envelope to determine the participant's group allocation and dispense the appropriate IV medications. Both envelopes will then be sealed and place in the participants chart. The envelopes will only be opened in the case of emergency unblinding or by study staff for data entry at a later date.

The Procedure:

The participant will undergo her procedure with the pain control regimen based on the randomization. The anesthetist will maintain a drug administration log throughout the procedure, including the use of any reversal agents. The total amounts of drugs mixed, used and wasted will be recorded in this log. Only the anesthetist will have access to this log in order to maintain blinding. It will be sealed and kept in the participants chart after the procedure is complete. It will only be opened if emergency unblinding is required or by research staff for data entry at a later date.

Once the procedure is complete, the nurse and/or surgeon will administer the immediate post-operative pain assessment. The surgeon will record their assessment of intra-operative pain management and their guess as to group assignment. Any adverse events or medication side effects during the procedure will be recorded by the clinical team (nurses and surgeons).

The Recovery Room:

In the recovery room, the clinical team (nurses and surgeons) will record any side effects or adverse events. Length of stay in recovery will be recorded in minutes by the nursing staff. The participant will be administered a final pain assessment by nursing staff prior to discharge. The participant will also be given a self-administered questionnaire with questions about participant satisfaction, likelihood of using the same pain regimen at a future procedure, and their guess regarding their group assignment.

Follow-Up:

The participant will be contacted by a member of the research team within 2-4 weeks of the procedure. This will be done by telephone. The participant will be asked a series of questions relating to satisfaction, complications that may have arisen following discharge, the likelihood of using the same pain regimen at a future procedure, and their guess regarding their group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed first trimester pregnancy with an ultrasound showing a viable intrauterine pregnancy with a gestational age of less than 12 weeks since the last menstrual period
2. Unwanted pregnancy and consented to undergo a first trimester surgical abortion

Exclusion Criteria:

1. Age <18 years at the time of study enrollment
2. Known allergy or sensitivity to any of the medications used in the study
3. Any serious medical comorbidity that would make IV sedation contraindicated in an outpatient setting (ex. Heart disease, lung disease)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS Pain Score - Immediate Post-Procedure | Immediate Post-Procedure
  The primary outcome measure is mean difference in immediate post-operative pain measured by the visual analogue pain scale (VAS). The VAS is a validated tool for research in operative pain management. Using this scale, participants rate their current pain on a scale from 0 to 10 by drawing an "x" on the horizontal line. This line is 10cm long and the participant's pain level is measured using a ruler to the millimeter mark and translated to a score out of 100mm. If the "x" falls between millimeter marks on the ruler the reader will round up to the nearest mark.

SECONDARY OUTCOMES:
VAS Pain Score - Prior to Discharge | Prior to discharge from recovery room on day of procedure (typically within 1h post-procedure)
  This secondary outcome will post-operative pain prior to discharge measured by the visual analogue pain scale (VAS). The VAS is a validated tool for research in operative pain management. Using this scale, participants rate their current pain on a scale from 0 to 10 by drawing an "x" on the horizontal line. This line is 10cm long and the participant's pain level is measured using a ruler to the millimeter mark and translated to a score out of 100mm. If the "x" falls between millimeter marks on the ruler the reader will round up to the nearest mark.
Length of Stay in Recovery | Day of Procedure
  Length of stay in recovery in minutes from transfer from the procedure room till discharge.
Satisfaction with Pain Control - Prior to Discharge | Prior to discharge from recovery room on day of procedure (typically within 1h post-procedure)
  Satisfaction with pain control will be assessed using a 5-point Likert scale. 1 is the worst score and 5 is the best.
Medication Side Effects | Prior to discharge from recovery room on day of procedure (typically within 1h post-procedure)
  Medication side effects from administration till discharge as reported by the care providers and nurses.
Provider Assessment of Intra-Operative Pain Management | Intra-Operative
  Provider assessment of intra-operative pain will be reported using a 5-point Likert scale. 1 is the worst score and 5 is the best.
Wong-Baker Faces Pain Score - Immediate Post-Procedure | Immediate Post-Procedure
  Pain score will immediate post-procedure will also be reported using the Wong-Baker Faces Pain Rating Scale.
Wong-Baker Faces Pain Score - Prior to Discharge | Prior to discharge from recovery room on day of procedure (typically within 1h post-procedure)
  Pain score will prior to discharge will also be reported using the Wong-Baker Faces Pain Rating Scale.
Pain Control After Discharge | 2-4 weeks post-procedure
  Pain control after discharge will be assessed via telephone questionnaire using a 5-point Likert scale. 1 is the worst score and 5 is the best.
Satisfaction with Pain Control After Discharge | 2-4 weeks post-procedure
  Satisfaction with pain control after discharge will be assessed via telephone questionnaire using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Bussiere-Cote, MD, Principal Investigator — Queen's University; Ashley Waddington, MD, MPA, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Induced abortions reported in Canada in 2016. Ottawa: Canadian Institute for Health Information; 2018. Available at: https://www.cihi.ca/en/induced-abortions-reported-in-canada-in-2016. Accessed on July 29, 2018.
- [Background] Costescu D, Guilbert E. No. 360-Induced Abortion: Surgical Abortion and Second Trimester Medical Methods. J Obstet Gynaecol Can. 2018 Jun;40(6):750-783. doi: 10.1016/j.jogc.2017.12.010. PMID 29861084
- [Background] Allen RH, Fitzmaurice G, Lifford KL, Lasic M, Goldberg AB. Oral compared with intravenous sedation for first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):276-83. doi: 10.1097/AOG.0b013e3181938758. PMID 19155895
- [Background] Agostini A, Maruani J, Roblin P, Champion J, Cravello L, Gamerre M. A double-blind, randomized controlled trial of the use of a 50:50 mixture of nitrous oxide/oxygen in legal abortions. Contraception. 2012 Jul;86(1):79-83. doi: 10.1016/j.contraception.2011.11.015. Epub 2012 Jan 20. PMID 22264664
- [Background] Kan AS, Caves N, Wong SY, Ng EH, Ho PC. A double-blind, randomized controlled trial on the use of a 50:50 mixture of nitrous oxide/oxygen in pain relief during suction evacuation for the first trimester pregnancy termination. Hum Reprod. 2006 Oct;21(10):2606-11. doi: 10.1093/humrep/del234. Epub 2006 Jun 21. PMID 16790607
- [Background] Strayer RJ, Nelson LS. Adverse events associated with ketamine for procedural sedation in adults. Am J Emerg Med. 2008 Nov;26(9):985-1028. doi: 10.1016/j.ajem.2007.12.005. PMID 19091264
- [Background] Galloon S. Ketamine for dilatation and curettage. Can Anaesth Soc J. 1971 Nov;18(6):600-13. doi: 10.1007/BF03026180. No abstract available. PMID 5119802
- [Background] Hejja P, Galloon S. A consideration of ketamine dreams. Can Anaesth Soc J. 1975 Jan;22(1):100-5. doi: 10.1007/BF03004825. PMID 1109698
- [Background] Erbguth PH, Reiman B, Klein RL. The influence of chlorpromazine, diazepam, and droperidol on emergence from ketamine. Anesth Analg. 1972 Sep-Oct;51(5):693-700. No abstract available. PMID 4560720
- [Background] Hervey WH, Hustead RF. Ketamine for dilatation and currettage procedures: patient acceptance. Anesth Analg. 1972 Jul-Aug;51(4):647-55. PMID 5064798
- [Background] Krestow M. The effect of post-anaesthetic dreaming on patient acceptance of ketamine anaesthesia: a comparison with thiopentone-nitrous oxide anaesthesia. Can Anaesth Soc J. 1974 Jul;21(4):385-9. doi: 10.1007/BF03006072. No abstract available. PMID 4836917
- [Background] Freuchen I, Ostergaard J, Kuhl JB, Mikkelsen BO. Reduction of psychotomimetic side effects of Ketalar (ketamine) by Rohypnol (flunitrazepam). A randomized, double-blind trial. Acta Anaesthesiol Scand. 1976;20(2):97-103. doi: 10.1111/j.1399-6576.1976.tb05015.x. PMID 7095
- [Background] Coad NR, Mills PJ, Verma R, Ramasubramanian R. Evaluation of blood loss during suction termination of pregnancy: ketamine compared with methohexitone. Acta Anaesthesiol Scand. 1986 Apr;30(3):253-5. doi: 10.1111/j.1399-6576.1986.tb02407.x. PMID 3739583
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman AB. Pain control in first-trimester surgical abortion: a systematic review of randomized controlled trials. Contraception. 2010 May;81(5):372-88. doi: 10.1016/j.contraception.2009.12.008. Epub 2010 Jan 27. PMID 20399943
- [Background] Godwin SA, Burton JH, Gerardo CJ, Hatten BW, Mace SE, Silvers SM, Fesmire FM; American College of Emergency Physicians. Clinical policy: procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2014 Feb;63(2):247-58.e18. doi: 10.1016/j.annemergmed.2013.10.015. PMID 24438649
- [Background] Atkinson P, French J, Nice CA. Procedural sedation and analgesia for adults in the emergency department. BMJ. 2014 May 8;348:g2965. doi: 10.1136/bmj.g2965. No abstract available. PMID 24812113
- [Background] Green SM, Roback MG, Kennedy RM, Krauss B. Clinical practice guideline for emergency department ketamine dissociative sedation: 2011 update. Ann Emerg Med. 2011 May;57(5):449-61. doi: 10.1016/j.annemergmed.2010.11.030. Epub 2011 Jan 21. PMID 21256625
- [Background] Newton A, Fitton L. Intravenous ketamine for adult procedural sedation in the emergency department: a prospective cohort study. Emerg Med J. 2008 Aug;25(8):498-501. doi: 10.1136/emj.2007.053421. PMID 18660398
- [Background] Coralic Z, Sawe HR, Mfinanga JA, Cortez A, Koehl J, Siroker H, Reynolds TA. Ketamine procedural sedation in the emergency department of an urban tertiary hospital in Dar es Salaam, Tanzania. Emerg Med J. 2018 Apr;35(4):214-219. doi: 10.1136/emermed-2017-206974. Epub 2018 Jan 22. PMID 29358491
- [Background] Bisanzo M, Nichols K, Hammerstedt H, Dreifuss B, Nelson SW, Chamberlain S, Kyomugisha F, Noble A, Arthur A, Thomas S. Nurse-administered ketamine sedation in an emergency department in rural Uganda. Ann Emerg Med. 2012 Apr;59(4):268-75. doi: 10.1016/j.annemergmed.2011.11.004. Epub 2011 Dec 9. PMID 22169331
- [Background] Sacchetti A, Senula G, Strickland J, Dubin R. Procedural sedation in the community emergency department: initial results of the ProSCED registry. Acad Emerg Med. 2007 Jan;14(1):41-6. doi: 10.1197/j.aem.2006.05.023. Epub 2006 Aug 31. PMID 16946280
- [Background] Allen RH, Singh R. Society of Family Planning clinical guidelines pain control in surgical abortion part 1 - local anesthesia and minimal sedation. Contraception. 2018 Jun;97(6):471-477. doi: 10.1016/j.contraception.2018.01.014. Epub 2018 Jan 31. PMID 29407363